CLINICAL TRIAL: NCT03446027
Title: A Multicenter Randomised Controlled Study: Does Neuromuscular Electrical Stimulation Improve the Absolute Walking Distance in Patients With Intermittent Claudication (NESIC) Compared to Best Available Treatment?
Brief Title: Does Neuromuscular Electrical Stimulation Improve the Absolute Walking Distance in Patients With Intermittent Claudication Compared to Best Available Treatment?
Acronym: NESIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17HH4216
Record Dates: First submitted 2018-01-08; First posted 2018-02-26 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Intermittent Claudication; Peripheral Vascular Diseases
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): There will be no change to the local site standard of care for patients with IC attributed to participation in this trial. Those sites with Supervised Exercise Therapy (SET) will continue to provide this intervention as per their normal standard of care and locally agreed protocol.
- Device (Experimental): Local therapy + Neuromuscular Electrical Stimulation (NMES)
  Interventions: Device: NMES

INTERVENTIONS:
Device: NMES — NMES device to be used for up to 3 hours daily in 30 minute sessions for 3 months.
  Arms: Device

SUMMARY:
Intermittent claudication (IC) is caused by a blockage in the artery of the leg, causing muscle pain. Although some evidence of the efficacy of neuromuscular electrical stimulation (NMES) in the management of patients with IC exists, further high quality research is required. This proposed study is vital to identify the contribution of clinical change using NMES, compared to the current gold standard recommended practice of supervised exercise therapy (SET) and, actual standard of care offered in the majority of the UK and Ireland, including best medical therapy (BMT). The device is expected to increase the walking distance in patients with intermittent claudication (IC), and therefore have a benefit on the same when provided in addition to supervised exercise programmes. It is also expected to cause a reduction in pain symptoms and reduced likelihood of major intervention in late stage peripheral arterial disease (PAD). The principal research objective is to assess the clinical efficacy of a neuromuscular electrical stimulation (NMES) device as an adjunct to the local standard care that is available at the study randomisation sites, in order to improve walking distance in patients with intermittent claudication (IC).

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent
* Aged 18 or above
* Positive Edinburgh Claudication Questionnaire
* ABPI <0.9 OR positive stress test (fall in ankle pressure >30mmHg, 40 secs post 1 min treadmill at 10% gradient, 4 km/h)

Exclusion Criteria:

* Severe IC requiring invasive intervention as determined by the treating clinician
* Critical limb Ischaemia as defined by the European Consensus Document
* Co-morbid disease prohibiting walking on a treadmill or taking part in supervised exercise therapy.
* Popliteal entrapment syndrome
* Commenced vascular symptom specific medication in previous 6 months e.g. naftidrofuryl oxalate, cilostazol
* Pregnancy
* Any implanted electronic, cardiac or defibrillator device
* Acute deep vein thrombosis
* Broken or bleeding skin including leg ulceration
* Peripheral neuropathy
* Recent lower limb injury or lower back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Davies, Principal Investigator — Chief Investigator
Locations (11):
- United Kingdom (11):
  - The Royal Bournemouth & Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - North Bristol NHS Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Dorset County Hospital NHS Foundation Trust, Dorchester
  - Hull and East Yorkshire Hospitals NHS Foundation Trust, Hull
  - Imperial College Healthcare NHS Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Taunton and Somerset NHS Foundation Trust, Taunton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Device
Started | 102 | 98
Completed | 78 | 80
Not Completed | 24 | 18

BASELINE CHARACTERISTICS:
Population: Baseline analysis including all patents randomised minus those removed post-randomisation due to screen failures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Device | Total
Number analyzed (Participants) | 98 | 92 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.44 (9.44) | 68.17 (8.84) | 67.79 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 70 | 70 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 90 | 87 | 177
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.63 (6.66) | 28.10 (5.12) | 28.37 (5.95)
Smoking status [Number; unit: participants]
  Current smoker | 34 | 22 | 56
  Former smoker | 58 | 64 | 122
  Never | 6 | 6 | 12
Medical history [Number; unit: participants]
  Hypertension | 63 | 65 | 128
  Stroke | 9 | 9 | 18
  Heart attack | 17 | 15 | 32
  High cholesterol | 64 | 68 | 132
  Angina | 13 | 10 | 23
  Diabetes | 26 | 21 | 47
  Bypass revascularisation | 12 | 5 | 17
  Angio revascularisation | 25 | 14 | 39
Medication [Number; unit: participants]
  Antiplatelets | 79 | 75 | 154
  Lipid modification therapy | 81 | 80 | 161
  Anticoagulant | 15 | 10 | 25
  Antihypertensives | 65 | 66 | 131
Retired [Number; unit: participants]
  Yes | 69 | 68 | 137
  No | 29 | 24 | 53
Work status [Number; unit: participants] — Only people who are not retired are reported Population: Only participants not retired were assessed and are reported for this Baseline Measure
  participants
    Higher managerial and professional occupations: number analyzed (Participants) | 29 | 24 | 53
    Higher managerial and professional occupations | 5 | 3 | 8
    Intermediate occupations (e.g. clerical, sales, service): number analyzed (Participants) | 29 | 24 | 53
    Intermediate occupations (e.g. clerical, sales, service) | 4 | 5 | 9
    Lower managerial and professional occupations: number analyzed (Participants) | 29 | 24 | 53
    Lower managerial and professional occupations | 1 | 8 | 9
    Lower supervisory and technical occupations: number analyzed (Participants) | 29 | 24 | 53
    Lower supervisory and technical occupations | 1 | 1 | 2
    Never worked or long-term unemployed: number analyzed (Participants) | 29 | 24 | 53
    Never worked or long-term unemployed | 7 | 2 | 9
    Routine occupations: number analyzed (Participants) | 29 | 24 | 53
    Routine occupations | 6 | 4 | 10
    Semi-routine occupations: number analyzed (Participants) | 29 | 24 | 53
    Semi-routine occupations | 2 | 1 | 3
    Small employers and own account workers: number analyzed (Participants) | 29 | 24 | 53
    Small employers and own account workers | 3 | 0 | 3
Performance limited due to intermittent claudication [Number; unit: participants] — Population: Only participants not retired were assessed and are reported for this Baseline Measure
  participants
    A little: number analyzed (Participants) | 29 | 24 | 53
    A little | 9 | 7 | 16
    A lot: number analyzed (Participants) | 29 | 24 | 53
    A lot | 4 | 3 | 7
    Not at all: number analyzed (Participants) | 29 | 24 | 53
    Not at all | 9 | 12 | 21
    Missing: number analyzed (Participants) | 29 | 24 | 53
    Missing | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Absolute Walking Distance (AWD) at 3 Months Between the Two Treatment Groups
Description: Measured by treadmill testing. Absolute walking distance in meters at baseline and 3 months
Time Frame: 3 months
Population: Control group includes both BMT and BMT + SET and the treatment group includes NMES + BMT and NMES + BMT + SET Included participants with both baseline and 3 month treadmill data.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Control: Control: Local Available Exercise Therapy (BMT and BMT+SET) as reference category. Treatment: BMT+NMES and BMT+SET+NMES
- Device: NMES + EA and NMES+EA+SET
Arm/Group | Control | Device
Number analyzed (Participants) | 98 | 92
Meters
  Baseline | 220.12 (148.27) | 242.97 (187.08)
  3 months | 327.74 (222.65) | 370.38 (251.38)
Statistical Analysis 1: Comparison: Control vs Device; Right censored Tobit regression model for AWD at 3 months for the ITT population. Difference between arms (between baseline and 3 months) - the primary analysis estimates the difference in the AWD at 3 months between the two treatment groups control vs. device. Control group includes both BMT and BMT + SET and the treatment group includes NMES + BMT and NMES + BMT + SET Included participants with both baseline and 3 month treadmill data; Test type: Other — Prespecified Tobit Regression mode: the model included the AWD baseline measurement, a treatment indicator and the type of centre (SET versus non-SET) as covariates. As the data collected for AWD showed a right-skewed distribution, a square root transformation was used to normalise the data and used for the regression Tobit model. This resulted in the unit of measure being "units" rather than meters; p = 0.28, Tobit Regression; square root transformation = 0.835, 95% CI 2-sided [-0.674 to 2.343]

2. Secondary Outcome: Difference in the Initial Claudication Distance (ICD) at 3 Months Between the Two Treatment Groups
Description: Measured by treadmill testing. ICD in meters at baseline and 3 months
Time Frame: 3 months
Population: Included participants with both baseline and 3 month treadmill data. Control group includes both BMT and BMT + SET and the treatment group includes NMES + BMT and NMES + BMT + SET
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Control: Control: Local Available Exercise Therapy (BMT and BMT+SET) as reference category.
- Device: BMT+NMES and BMT+SET+NMES
Arm/Group | Control | Device
Number analyzed (Participants) | 98 | 92
Meters
  Baseline | 99.10 (77.06) | 105.79 (106.27)
  3 months: number analyzed (Participants) | 80 | 80
  3 months | 179.73 (147.03) | 211.45 (181.83)
Statistical Analysis 1: Comparison: Control vs Device; Test type: Other — Right censored, Tobit Regression model to assess the effects of baseline characteristics for ICD at 3 months for the ITT Population. This resulted in the unit of measure being "units" and not meters. Included participants with both baseline and 3 month treadmill data. Calculation between arms - estimates the difference in the ICD at 3 months between the two treatment groups. Control group includes both BMT and BMT + SET and the treatment group includes NMES + BMT and NMES + BMT + SET; p = 0.23, Right censored, Tobit Regression; square root transformation = 0.972, 95% CI 2-sided [-0.600 to 2.546]

3. Secondary Outcome: Quality of Life - Intermittent Claudication Questionnaire (ICQ)
Description: Patient questionnaire. Used to assess change in disease-specific QoL.
Time Frame: Baseline, 3 months, 6 months, 12 months
Population: Scores on the Intermittent Claudication Questionnaire range from 0 to 100, with higher scores indicating worse health related to intermittent claudication.
  Includes all participants that completed the ICQ questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Device
Number analyzed (Participants) | 94 | 90
score on a scale
  Baseline | 45.92 (13.09) | 41.98 (13.26)
  3 months | 41.33 (14.52) | 36.55 (13.86)
  6 months | 39.27 (14.51) | 35.20 (15.07)
  12 months | 36.21 (16.45) | 36.99 (17.38)

4. Secondary Outcome: Quality of Life - EuroQoL 5D (EQ5D) Health Scale
Description: Patient questionnaire. Used to assess the generic QoL and will allow economic assessment based on intervention and score improvement.
Time Frame: Baseline, 3 month, 6 month and 12 months
Population: Scores on the EuroQol Group 5-Dimension 5-Level questionnaire (EQ-5D-5L) health scale (a visual-analogue scale) range from 0 to 100, with higher scores indicating better health.
  Includes all participants that completed the EQ-5D-5L questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Device
Number analyzed (Participants) | 97 | 91
score on a scale
  Baseline | 45.92 (13.09) | 41.98 (13.26)
  3 months | 41.33 (14.52) | 36.55 (13.86)
  6 months | 39.27 (14.51) | 35.20 (15.07)
  12 months | 36.21 (16.45) | 36.99 (17.38)

5. Secondary Outcome: Quality of Life Short Form 36 (SF-36) Physical Component Summary
Description: as for outcome 4
Time Frame: Baseline, 3 month, 6 month and 12 months
Population: Scores on the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Physical Component Summary and Mental Component Summary range from 1 to 100, with higher scores indicating better quality of life.
  Includes all participants that completed the SF-36 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Device
Number analyzed (Participants) | 95 | 91
score on a scale
  Baseline | 36.14 (7.90) | 35.71 (8.22)
  3 months | 37.42 (8.48) | 38.80 (8.87)
  6 months | 37.62 (9.85) | 39.47 (9.74)
  12 months | 39.46 (9.40) | 38.16 (9.98)

6. Secondary Outcome: Haemodynamic Assessment - Duplex Ultrasonography - Difference in Volume Flow Between Baseline and 3 Months
Description: Using an arterial ultrasound probe and pre-set volume flow algorithms on a duplex ultrasound machine, flow within the common femoral artery (CFA), of the most affected limb, will be measured, approximately 5cm below the mid-inguinal point at the groin. Measures include volume flow (VF, cc/min) to assess whether using the device increases this measurement.
Time Frame: 3 months
Population: Includes all participants that had a volume flow measurement at baseline and 3 months
Measure: Mean (Standard Deviation); unit: cc/min
Groups:
- Device: Treatment: BMT+NMES and BMT+SET+NMES
Arm/Group | Control | Device
Number analyzed (Participants) | 87 | 80
cc/min
  Baseline | 296.89 (198.40) | 300.06 (155.10)
  3 months: number analyzed (Participants) | 71 | 71
  3 months | 280.96 (179.03) | 296.77 (146.30)
Statistical Analysis 1: Comparison: Control vs Device; Test type: Other — Linear Regression Model for Duplex ultrasonography (Volume flow - measured in one leg) at 3 months for the ITT population. Difference (calculation) between the two groups and not per arm (control vs treatment). Unit of measure is "Units" due to the use of a linear regression model rather than cc/min; p = 0.516, Regression, Linear; Linear regression = 0.483, 95% CI 2-sided [-0.984 to 1.950]

7. Secondary Outcome: Haemodynamic Assessment - Laser Doppler Flowmetry (LDF) - Difference in Blood Flux Between Baseline and 12 Months
Description: The single fibre laser optical probe of the LDF machine will be positioned on the dorsal aspect of the foot using single use adhesive pads. Flux, as a measure of superficial skin blood flow will be measured to assess whether using the device increases this measurement.
Time Frame: Baseline, 3 month, 6 month and 12 months
Population: ANCOVA model for changes in Laser Doppler Flowmetry (blood flux - measured in one leg) between baseline and follow up periods (3, 6 and 12 months) for the ITT population.
  Includes all participants that completed the LDF assessment. Blood flux is unitless. Difference between the two groups (control vs device).
Measure: Mean (Standard Deviation); unit: Unitless
Groups:
- Treatment: BMT+NMES and BMT+SET+NMES
- Control: BMT and BMT+SET
Arm/Group | Treatment | Control
Number analyzed (Participants) | 90 | 96
Unitless
  Baseline | 2.61 (0.58) | 2.38 (0.56)
  3 months | 2.79 (0.69) | 2.30 (0.65)
  6 months | 2.49 (0.57) | 2.50 (0.62)
  12 months | 2.64 (0.61) | 2.53 (0.56)

8. Secondary Outcome: Haemodynamic Assessment - Difference in Ankle Brachial Pressure Index (ABPI) - Left - Between Baseline and 12 Months
Description: The brachial blood pressure from the right arm using a manual blood pressure monitor cuff and Doppler will be recorded after 5 minutes of resting supine on a couch. The systolic blood pressure of the anterior tibial artery and posterior tibial artery at the ankle will also be recorded using the cuff and Dopplermethod. The ratio of the systolic brachial and ankle pressures will form the ABPI measurement.
Time Frame: Baseline, 3 month, 6 month and 12 months
Population: Linear mixed model for changes in the transformed log Left Ankle Brachial Pressure Index (ABPI) between baseline and follow up periods (3, 6 and 12 months) for the ITT population.
  Calculation between groups - assesses the difference between the two treatment groups between baseline and 12 months.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Control | Device
Number analyzed (Participants) | 97 | 90
Ratio
  Baseline | 0.76 (0.21) | 0.72 (0.18)
  3 months: number analyzed (Participants) | 79 | 81
  3 months | 0.74 (0.23) | 0.72 (0.21)
  6 months: number analyzed (Participants) | 67 | 71
  6 months | 0.77 (0.22) | 0.74 (0.2)
  12 months: number analyzed (Participants) | 64 | 53
  12 months | 0.79 (0.23) | 0.74 (0.22)

9. Secondary Outcome: Health Economic Assessment
Description: The economic analyses will compare local therapy (supervised exercise therapy (SET) or exercise advice (EA) only) versus the intervention (local therapy + Neuromuscular Electrical Stimulation, NMES) in patients with Intermittent Claudication. The analyses will be based on a (i) patient level in-trial cost-effectiveness analysis, (ii) a decision model and (iii) budget impact assessment. The in-trial analysis will calculate quality-adjusted life years (QALYs) over the one year time horizon of the trial.
Time Frame: Baseline, 3 month, 6 month and 12 months
Population: All randomised patients (except screen failures)
Measure: Mean (95% Confidence Interval); unit: QALY
Arm/Group | Treatment | Control
Number analyzed (Participants) | 98 | 102
QALY | 0.6459 [0.6032 to 0.6886] | 0.6355 [0.5992 to 0.6718]

10. Secondary Outcome: Compliance With Interventions - Exercise Advice (EA)
Description: Comparison of compliance with exercise advice as per local standard of care.
Time Frame: 3 months
Population: EA (part of BMT): compliant if completed 75% or more of recommended level of EA (75% of minutes performing exercises recommended by centre).
  Data for this Outcome Measure was pre-specified to be collected and assessed as a single group irrespective of intervention Arm/Group.
Measure: Count of Participants; unit: Participants
Groups:
- Compliance to Exercise Advice: Exercise advice (EA) (part of best medical therapy): compliant if completed 75% or more of recommended level of EA (75% of minutes performing exercises recommended by centre).
Arm/Group | Compliance to Exercise Advice
Number analyzed (Participants) | 190
Participants
  Complier | 99
  Non-complier | 52
  Missing | 39

11. Secondary Outcome: Device Experience Questionnaire - Ease of Use
Description: To report ease of device use and suggest any developments.
Time Frame: 3 months
Population: Participants asked to rate ease of use of device. 5 point scale from 1 (very easy) to 5 (very difficult) Includes all participants that were in the control arm and completed the device experience questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- Device Arm: Reduces leg pain
Arm/Group | Device Arm
Number analyzed (Participants) | 88
Participants
  1 Very easy | 77
  2 | 6
  3 | 1
  4 | 0
  5 Very difficult | 0
  Missing | 4

12. Secondary Outcome: Quality of Life - EuroQoL 5D (EQ5D) Health Index
Description: as for outcome 4
Time Frame: Baseline, 3 months, 6 months, 12 months
Population: Score on the EQ-5D-5L health index range from 0 to 100, with higher scores indicating better health. The EQ-5D-5L health index was calculated with the value set for England.
  Includes all participants that completed the EuroQoL 5D (EQ5D) Health Index.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Device
Number analyzed (Participants) | 97 | 91
score on a scale
  Baseline | 69.61 (17.69) | 69.73 (18.03)
  3 months | 66.11 (21.09) | 74.02 (15.13)
  6 months | 68.36 (20.85) | 73.13 (19.32)
  12 months | 68.03 (19.61) | 70.40 (20.98)

13. Secondary Outcome: Quality of Life Short Form 36 (SF-36) Mental Component Summary
Description: as for outcome 4
Time Frame: Baseline, 3 months, 6 months, 12 months
Population: Scores on the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Physical Component Summary and Mental Component Summary range from 1 to 100, with higher scores indicating better quality of life.
  Includes all participants that completed the SF-36 Mental Component Summary.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Device
Number analyzed (Participants) | 95 | 91
score on a scale
  Baseline | 49.75 (12.47) | 52.06 (11.61)
  3 months | 48.24 (13.15) | 52.99 (10.05)
  6 months | 49.09 (10.90) | 52.79 (10.73)
  12 months | 48.90 (12.24) | 52.62 (11.68)

14. Secondary Outcome: Haemodynamic Assessment - Duplex Ultrasonography - Difference in Time Average Mean Velocity Between Baseline and 3 Months
Description: Using an arterial ultrasound probe and pre-set volume flow algorithms on a duplex ultrasound machine, flow within the common femoral artery (CFA), of the most affected limb, will be measured, approximately 5cm below the mid-inguinal point at the groin. Measures include time-averaged mean volume (TAMV, cm/s) to assess whether using the device increases this measurement.
Time Frame: 3 months
Population: Linear Regression Model for Duplex ultrasonography (TAMV - measured in one leg) at 3 months for the ITT population.
  Difference (calculation) between the two groups (control and treatment) and not per arm.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Control | Device
Number analyzed (Participants) | 89 | 81
cm/s
  Baseline | 11.28 (5.64) | 12.23 (6.47)
  3 months: number analyzed (Participants) | 72 | 71
  3 months | 11.78 (5.77) | 12.47 (5.39)

15. Secondary Outcome: Haemodynamic Assessment - Difference in Ankle Brachial Pressure Index (ABPI) - Right - Between Baseline and 12 Months
Description: as for outcome 8
Time Frame: Baseline, 3 months, 6 months and 12 months
Population: Linear mixed model1 for changes in the transformed log Right Ankle Brachial Pressure Index (ABPI) between baseline and follow up periods (3, 6 and 12 months) for the ITT population.
  Calculation between groups - assesses the difference between the two treatment groups between baseline and 12 months.
  Calculation between the two groups (control and treatment).
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Control | Device
Number analyzed (Participants) | 97 | 90
Ratio
  Baseline | 0.77 (0.22) | 0.76 (0.21)
  3 months | 0.78 (0.22) | 0.77 (0.21)
  6 months | 0.80 (0.28) | 0.76 (0.23)
  12 months | 0.79 (0.23) | 0.78 (0.21)

16. Secondary Outcome: Compliance With Interventions - Supervised Exercise Therapy (SET)
Description: Comparison of compliance with SET classes.
Time Frame: 3 months
Population: Participant's who attended SET programme.
Measure: Count of Participants; unit: Participants
Groups:
- Compliance to Supervised Exercise Therapy (SET): Compliant if attended 50% or more SET sessions held by centre
Arm/Group | Compliance to Supervised Exercise Therapy (SET)
Number analyzed (Participants) | 99
Participants
  Complier | 69
  Non-complier | 19
  Missing | 11

17. Secondary Outcome: Compliance With Interventions - Neuromuscular Electrical Stimulation (NMES)
Description: Compliance with NMES device. NMES compliance data collected from the data logger fitted to device and patient diary will be combined to report overall compliance.
Time Frame: 3 months
Population: NMES: compliant if completed 75% or more of recommended level of NMES usage.
Measure: Count of Participants; unit: Participants
Groups:
- Compliance to Neuromuscular Electrical Stimulation (NMES): NMES: compliant if completed 75% or more of recommended level of NMES usage.
Arm/Group | Compliance to Neuromuscular Electrical Stimulation (NMES)
Number analyzed (Participants) | 92
Participants
  Complier | 68
  Non-complier | 12
  Missing | 12

18. Secondary Outcome: Device Experience Questionnaire - Reduces Leg Pain
Description: To report ease of device use and suggest any developments.
Time Frame: 3 months
Population: Participants asked whether they thought the device reduced leg pain. 5-point scale from 1 (yes, a lot) to 5 (not at all).
  Includes all participants that were in the treatment (device) arm and that completed the device experience questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Arm
Number analyzed (Participants) | 88
Participants
  1-Yes, a lot | 14
  2 | 22
  3 | 26
  4 | 11
  5-Not at all | 11
  Missing | 4

19. Secondary Outcome: Device Experience Questionnaire - Increased Walk Distance
Description: To report ease of device use and suggest any developments.
Time Frame: 3 months
Population: Participants asked whether they thought the device increased walking distance. Includes all participants that were in the treatment (device) arm and that completed the device experience questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- Device Arm: Increased walk distance
Arm/Group | Device Arm
Number analyzed (Participants) | 88
Participants
  No | 8
  No change | 19
  Yes | 57
  Missing | 4

20. Secondary Outcome: Device Experience Questionnaire - Used as Instructed
Description: To report ease of device use and suggest any developments.
Time Frame: 3 months
Population: Participants asked whether they used the device as instructed. Includes all participants that were in the treatment (device) arm and that completed the device experience questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- Device Arm: Used as instructed
Arm/Group | Device Arm
Number analyzed (Participants) | 88
Participants
  No | 2
  Yes | 82
  Missing | 4

21. Secondary Outcome: Device Experience Questionnaire - Could Have Used More
Description: To report ease of device use and suggest any developments.
Time Frame: 3 months
Population: Participants asked whether they could have used the device more. Includes all participants that were in the treatment (device) arm and that completed the device experience questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- Device Arm: Could have used more
Arm/Group | Device Arm
Number analyzed (Participants) | 88
Participants
  No | 28
  Yes | 56
  Missing | 4

22. Secondary Outcome: Device Experience Questionnaire - Used After Treatment
Description: To report ease of device use and suggest any developments.
Time Frame: 3 months
Population: Participants asked whether they used the device following the 3 month treatment period. 5-point scale from 1 (Yes, a lot) to 5 (not at all).
  Includes all participants that were in the treatment (device) arm and that completed the device experience questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- Device Arm: Used after treatment
Arm/Group | Device Arm
Number analyzed (Participants) | 88
Participants
  1-Yes, a lot | 51
  2 | 13
  3 | 16
  4 | 0
  5-Not at all | 4
  Missing | 4

23. Other Pre Specified Outcome: Sub-group Analysis 1 - Difference in Absolute Walking Difference Between Baseline and 3 Months SET Sites vs Non-SET Sites
Description: Subgroup analysis 1: Right censored Tobit regression model for AWD at 3 months to assess the effects SET sites vs non-SET sites (NMES+SET+BMT & SET+BMT vs NMES+BMT & BMT).
Time Frame: 3 months
Population: Subgroup analysis 1: Treatment effect in SET sites vs non-SET sites (NMES+SET+BMT & SET+BMT vs NMES+BMT & BMT).
  Right censored Tobit regression model for AWD at 3 months to assess the effects of SET vs non-SET (subgroup1) for the ITT population (N=160).
  Subgroup1 (Non-SET) as reference category. Between group calculation (not per arm). Unit of measure is "Units" as a square root transformation was used to normalise the data and used for the Regression Tobit model, rather than meters.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Treatment Effect in SET Sites vs Non-SET Sites: Subgroup analysis 1: Treatment effect in SET sites vs non-SET sites (NMES+SET+BMT & SET+BMT vs NMES+BMT & BMT).
Arm/Group | Treatment Effect in SET Sites vs Non-SET Sites
Number analyzed (Participants) | 160
Units | 3.205 [1.689 to 4.720]

24. Other Pre Specified Outcome: Sub-group Analysis 2 - Difference in Absolute Walking Difference Between Baseline and 3 Months (NMES+SET+BMT vs SET+BMT)
Description: Subgroup analysis 2: Right censored Tobit Regression model for AWD at 3 months to assess the effects of NMES in the SET sites (NMES+SET+BMT vs SET+BMT).
Time Frame: 3 months
Population: Subgroup analysis 2: Treatment effect of NMES in the SET sites (NMES+SET+BMT vs SET+BMT).
  Right censored Tobit Regression model for AWD at 3 months to assess the effects of EA+SET+NMES vs EA+SET (subgroup2) for the ITT population (N=90) Subgroup2 (BMT + SET) as reference category. Between group calculation (not per arm). Unit of measure is "Units" as a square root transformation was used to normalise the data and used for the Regression Tobit model, rather than meters.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Treatment Effect of NMES in the SET Sites: Subgroup analysis 2: Treatment effect of NMES in the SET sites (NMES+SET+BMT vs SET+BMT).
Arm/Group | Treatment Effect of NMES in the SET Sites
Number analyzed (Participants) | 90
Units | 1.724 [-0.560 to 4.008]

25. Other Pre Specified Outcome: Sub-group Analysis 3 - Difference in Absolute Walking Difference Between Baseline and 3 Months (NMES+BMT vs BMT)
Description: Subgroup analysis 3: Right censored Tobit regression model for the AWD at 3 months to assess the effects of NMES in the non-SET sites (NMES+BMT vs BMT).
Time Frame: 3 months
Population: Subgroup analysis 3: Treatment effect of NMES in the non-SET sites (NMES+BMT vs BMT).
  Right censored Tobit regression model for the AWD at 3 months to assess the effects of EA vs EA+NMES (subgroup3) for the ITT population (N=70) Subgroup3 (BMT) as reference category. Between group calculation (not per arm). Unit of measure is "Units" as a square root transformation was used to normalise the data and used for the Regression Tobit model, rather than meters.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Treatment Effect of NMES in the Non-SET Sites: Subgroup analysis 3: Treatment effect of NMES in the non-SET sites (NMES+BMT vs BMT). The sample size in this group is N=91 (n=46 in BMT and n=45 in BMT+NMES).
Arm/Group | Treatment Effect of NMES in the Non-SET Sites
Number analyzed (Participants) | 70
Units | -0.090 [-2.014 to 1.833]

26. Other Pre Specified Outcome: Sub-group Analysis 4 - Difference in Absolute Walking Difference Between Baseline and 3 Months (NMES+BMT vs. SET+BMT)
Description: Subgroup analysis 4: Right censored Tobit regression model for AWD at 3 months to assess the effects of (NMES+BMT) has a similar effect as (SET+BMT).
Time Frame: 3 months
Population: Subgroup analysis 4: Investigate if the treatment effect of (NMES+BMT) has a similar effect as (SET+BMT).
  Right censored Tobit regression model for AWD at 3 months to assess the effects of EA+SET vs EA+NMES (subgroup4) for the ITT population (N=88) Subgroup4 (BMT+SET) as reference category. Between group calculation (not per arm). Unit of measure is "Units" as a square root transformation was used to normalise the data and used for the Regression Tobit model, rather than meters.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Investigate if the Treatment Effect of (NMES+BMT) Has a Similar Effect as (SET+BMT): Subgroup analysis 4: Investigate if the treatment effect of (NMES+BMT) has a similar effect as (SET+BMT). The sample size in this group is N=97 (n=52 in BMT+SET and n=45 in BMT+NMES).
Arm/Group | Investigate if the Treatment Effect of (NMES+BMT) Has a Similar Effect as (SET+BMT)
Number analyzed (Participants) | 88
Units | -2.419 [-4.324 to -0.513]

27. Other Pre Specified Outcome: Sub-group Analysis 5 - Difference in Absolute Walking Difference Between Baseline and 3 Months (NMES+SET+BMT vs. NMES+BMT)
Description: Subgroup analysis 5: Determine if (NMES+SET+BMT) is more effective than (NMES+BMT).
Time Frame: 3 months
Population: Subgroup analysis 5: Determine if (NMES+SET+BMT) is more effective than (NMES+BMT).
  Right censored Tobit regression model for AWD at 3 months to assess the effects of EA+NMES vs EA+SET+NMES (subgroup5) for the ITT population (N=80).
  Subgroup5 (BMT+NMES) as reference category. Between group calculation (not per arm). Unit of measure is "Units" as a square root transformation was used to normalise the data and used for the Regression Tobit model, rather than meters.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Determine if (NMES+SET+BMT) is More Effective Than (NMES+BMT): Subgroup analysis 5: Determine if (NMES+SET+BMT) is more effective than (NMES+BMT). The sample size in this group is N=92 (n=45 in BMT+NMES and n=47 in BMT+SET+NMES).
Arm/Group | Determine if (NMES+SET+BMT) is More Effective Than (NMES+BMT)
Number analyzed (Participants) | 80
Units | 4.248 [2.229 to 6.268]

28. Post Hoc Outcome: Sub-group Analysis 6 - Difference in Absolute Walking Difference Between Baseline and 3 Months (BMT vs. NMES+SET+BMT)
Description: Subgroup analysis 6: Determine if (BMT) is more effective than (NMES+SET+BMT).
Time Frame: 3 months
Population: Subgroup analysis 6: Determine if (BMT) is more effective than (NMES+SET+BMT). Right censored Tobit regression model for AWD at 3 months to assess the effects of EA vs EA+SET+NMES (subgroup 6) for the ITT population (N=72) Subgroup6 (BMT+SET+NMES) as reference category. Between group calculation (not per arm). Unit of measure is "Units" as a square root transformation was used to normalise the data and used for the Regression Tobit model, rather than meters.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Determine if (BMT) is More Effective Than (NMES+SET+BMT): Subgroup analysis 6: Determine if (BMT) is more effective than (NMES+SET+BMT). The sample size in this group is N=93 (n=46 in BMT and n=47 in BMT+SET+NMES).
Arm/Group | Determine if (BMT) is More Effective Than (NMES+SET+BMT)
Number analyzed (Participants) | 93
Units | -4.098 [-6.560 to -1.636]

29. Post Hoc Outcome: Sub-group Analysis 7 - Difference in Absolute Walking Difference Between Baseline and 3 Months (BMT vs. BMT+SET)
Description: Subgroup analysis 7: Determine if (BMT) is more effective than (BMT+SET). The sample size in this group is N=80 (n=31 in BMT and n=49 in BMT+SET).
Time Frame: 3 months
Population: Subgroup analysis 7: Determine if BMT is more effective than BMT+SET. The sample size in this group is N=80 (n=31 in BMT and n=49 in BMT+SET). BMT as reference category.
  Right censored Tobit regression model for AWD at 3 months to assess the effects of BMT vs BMT+SET (subgroup 7) for the ITT population.
  Between group calculation (not per arm). Unit of measure is "Units" as a square root transformation was used to normalise the data and used for the Regression Tobit model, rather than meters.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Determine if (BMT) is More Effective Than (BMT+SET): Subgroup analysis 7: Determine if (BMT) is more effective than (BMT+SET). The sample size in this group is N=80 (n=31 in BMT and n=49 in BMT+SET).
Arm/Group | Determine if (BMT) is More Effective Than (BMT+SET)
Number analyzed (Participants) | 80
Units | 2.341 [0.054 to 4.629]

30. Post Hoc Outcome: Post-hoc: Difference in Absolute Walking Difference for Patients Who Walked a Short Distance at Baseline (Baseline to 3 Months)
Description: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a short distance at baseline in the ITT population (N=40). The AWD at baseline was divided into three strati: Short, Medium and Long distances (set at <25%, 25%-75% and >75% respectively) using the descriptive statistics - short distance defined as <100m.
Time Frame: 3 months
Population: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a short distance at baseline in the ITT population (N=40). Control: Local Available Exercise Therapy (BMT and BMT+SET) as reference category.
  Calculated between the two groups (control vs treatment) so not per arm.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Treatment Versus Control: Primary Outcome for Patients Who Walked a Short Distance at Baseline: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a short distance at baseline in the ITT population (N=40)
Arm/Group | Treatment Versus Control: Primary Outcome for Patients Who Walked a Short Distance at Baseline
Number analyzed (Participants) | 40
Units | 0.426 [-3.499 to 4.351]

31. Post Hoc Outcome: Post-hoc: Difference in Absolute Walking Difference for Patients Who Walked a Medium Distance at Baseline (Baseline to 3 Months)
Description: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a medium distance at baseline in the ITT population (N=80). The AWD at baseline was divided into three strati: Short, Medium and Long distances (set at <25%, 25%-75% and >75% respectively) using the descriptive statistics - medium distance defined as between 100m and 340m.
Time Frame: 3 months
Population: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a medium distance at baseline in the ITT population (N=80). Control: Local Available Exercise Therapy (BMT and BMT+SET) as reference category.
  Calculated between the two groups (control vs treatment) so not per arm.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Treatment Versus Control: Primary Outcome for Patients Who Walked a Medium Distance at Baseline: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a medium distance at baseline in the ITT population (N=80)
Arm/Group | Treatment Versus Control: Primary Outcome for Patients Who Walked a Medium Distance at Baseline
Number analyzed (Participants) | 80
Units | 0.215 [-1.805 to 2.235]

32. Post Hoc Outcome: Post-hoc: Difference in Absolute Walking Difference for Patients Who Walked a Long Distance at Baseline (Baseline to 3 Months)
Description: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a long distance at baseline in the ITT population (N=40). The AWD at baseline was divided into three strati: Short, Medium and Long distances (set at <25%, 25%-75% and >75% respectively) using the descriptive statistics - long distance defined as >340m.
Time Frame: 3 months
Population: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a long distance at baseline in the ITT population (N=40). Control: Local Available Exercise Therapy (BMT and BMT+SET) as reference category.
  Calculated between the two groups (control vs treatment) so not per arm.
Measure: Number (95% Confidence Interval); unit: Units
Groups:
- Treatment Versus Control: Primary Outcome for Patients Who Walked a Long Distance at Baseline: Right censored Tobit regression model for Absolute Walking Distance (AWD) at 3 months for patients who walked a long distance at baseline in the ITT population (N=40)
Arm/Group | Treatment Versus Control: Primary Outcome for Patients Who Walked a Long Distance at Baseline
Number analyzed (Participants) | 40
Units | 2.877 [0.506 to 5.248]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the full study duration (12 months).
Description: Same definitions as clinicaltrials.gov
Arm/Group | Control | Device
All-Cause Mortality (participants affected / at risk) | 2/102 | 2/98
Serious Adverse Events (participants affected / at risk) | 13/102 | 11/98
Other Adverse Events (participants affected / at risk) | 44/102 | 47/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=102) | Device (N=98)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Prostatic operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (2) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=102) | Device (N=98)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stricture of oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crying (General disorders) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 5 (7) | 4 (4)
Norovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (5) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (3)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Colporrhaphy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (1) | 2 (3)
Peripheral artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Suture removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (4)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
We did not stratify by baseline absolute walking distance AWD for the primary outcome analysis.

Only 160 patients had analysable primary outcome data due to missing treadmill data.

Absence of a sham device comparator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT03446027/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03446027/SAP_001.pdf